CLINICAL TRIAL: NCT05765045
Title: A Nursing Triage Protocol for Minor Orthopedic Traumata: the Effect on Flow Time, Quality of Care and Patient Satisfaction in an Emergency Department
Acronym: TRINU-RX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiteit Antwerpen (Other)
Collaborators: Heilig Hartziekenhuis, Mol (Unknown)
Responsible Party: Principal Investigator, Filip Haegdorens, Principal Investigator, Universiteit Antwerpen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: TRINU-RX
Record Dates: First submitted 2023-02-09; First posted 2023-03-13 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Trauma Injury
MeSH Terms: conditions — Accidental Injuries

STUDY DESIGN:
Intervention Model Description: Intervention group and control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nursing triage group (Experimental): Using a triage protocol for medical imaging conducted by a triage nurse in the emergency department
  Interventions: Diagnostic Test: Nursing triage protocol
- Regular care group (No Intervention): Regular triage in the emergency department

INTERVENTIONS:
Diagnostic Test: Nursing triage protocol — Medically approved and supervised standing order that allows trained ER nurses to start medical imaging (RX) for adult patients with minor traumata to the limbs.
  Arms: Nursing triage group

SUMMARY:
In 2019, nearly half of all hospital contacts in Belgium took place through the emergency department, and more than a third of patients arrived after an accident or trauma. In instances of overcrowding, patients with minor orthopedic injuries face prolonged waiting times. Previous studies have shown that implementing triage protocols for medical imaging conducted by a triage nurse can reduce the Total Length of Stay (TLOS) for this patient group.

This is a single-center, unblinded, randomized, controlled trial that aims to evaluate the impact of a nurse triage protocol on turnaround time (primary outcome), quality of care, and patient satisfaction. The study population consists of adults who present with minor orthopedic injuries below the elbow or knee and have an Emergency Severity Index (ESI) of 4 or 5. Participants are randomly assigned to either the 'nurse triage protocol' group (n=110) or the 'usual care' group (n=110).

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years old)
* ESI 4 or ESI 5 Recent trauma (< 10 days after trauma)
* Accidental trauma mechanism
* Trauma below the elbow (forearm, wrist, hand, finger)
* Trauma below the knee (lower leg, ankle, foot, toe)

Exclusion Criteria:

* ESI 1 or ESI 2 or ESI 3
* Return visit after previous emergency department contact for the same injury (e.g. increased pain, tight cast, ...)
* Trauma resulting from underlying somatic pathology (e.g. syncope, epileptic attack, vertigo, vasovagal collapse, ...)
* Atraumatic (pain) complaints (e.g. pain in the calf, toe, foot, wrist, ... without a clear trauma mechanism)
* Additional, non-orthopedic injuries (e.g. laceration, signs of cerebral commotion, ...)
* Pregnancy or a suspicion of pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2023-03-06 (Actual); Primary Completion 2023-04-23 (Actual); Study Completion 2023-04-23 (Actual)

PRIMARY OUTCOMES:
TLOS | 6-8 weeks
  Total length of stay

SECONDARY OUTCOMES:
Patient satisfaction | 6-8 weeks
  Patient satisfaction measured by a 10-point Likert scale at discharge using a questionnaire
Treatment efficiency | 6-8 weeks
  Measurement if the patient diagnosis and/or treatment was correctly initiated at the Emergency Department. Yes = no additional diagnosis or treatments were necessary; No = within 14 days after discharge a change in treatment or new diagnosis was done. Data will be collected using the hospital's patient records or by calling patients if no information is found in the record.

CONTACTS AND LOCATIONS:
Overall Officials: Filip Haegdorens, PhD, Principal Investigator — Universiteit Antwerpen
Locations (1):
- University of Antwerp, Wilrijk, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No